CLINICAL TRIAL: NCT07084597
Title: Effect of Vitamin D3 Supplementation on Cardiac Autonomic Nerve Function in Male
Brief Title: Effect of Vitamin D3 Supplementation on Cardiac Autonomic Nerve Function in Male Parkinson's Disease Patients With Hypovitaminosis D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bangladesh Medical University (Other)
Responsible Party: Principal Investigator, Jobayda Binte Rahmatullah, MD Resident, Bangladesh Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5600
Record Dates: First submitted 2025-07-17; First posted 2025-07-24 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease
Keywords: Vitamin D3; HRV; Hypovitaminosis D; Parkinson disease
MeSH Terms: conditions — Parkinson Disease; Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: 15 male Parkinson's disease patients with hypovitaminosis D will be enrolled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 15 male Parkinson's disease patients (Experimental): 15 male Parkinson's disease patients with hypovitaminosis D will be enrolled. They will be supplemented with vitamin D orally 50,000 IU/weeks for 8 weeks
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — Vitamin D ,50000 IU/week will be given for 8 consecutive weeks

SUMMARY:
The goal of this clinical trial is to see the effect of vitamin D3 supplementation on cardiac autonomic nerve function in male Parkinson's disease patients with hypovitaminosis D

Main questions it aims to answer are:

1. Does vitamin D improves heart rate variability(HRV) in male Parkinson's disease patients ?
2. Does vitamin D improves cardiac autonomic nerve function in male Parkinson's disease patients ? It is a self control trial. Vitamin D3 deficient Parkinson's disease participants will

a. undergo through baseline HRV test b. Then they will take vitamin D3 capsule 50000 IU once in a week for 8 consecutive weeks c. Then after intervention with vitamin D supplementation post interventional HRV will be done.

Researcher will compare pre intervention(pre test) and post intervention(post test) value of HRV

DETAILED DESCRIPTION:
In Parkinson's disease , there is a shifting of autonomic nerve function towards sympathetic dominance and Heart rate variability decrease. Reduced heart rate variability can be detected by Heart rate variability(HRV) testing.

In Parkinson's disease deposition of Lewy bodies (due to accumulation of alpha- synuclein protein ) causes degeneration of dopaminergic neuron. Parasympathetic nerve results from vagus nerve atrophy and simultaneous sympathetic denervation results in decrease HRV.

Hypovitaminosis D is commonly associated with Parkinson's disease due to alteration of gastrointestinal function, progressive skin atrophy, lack of mobilization, lack of sun exposure.

Vitamin D3 act as neuroprotective hormone and plays role in autonomic nervous system regulation and maintaining balance between sympathetic and parasympathetic nervous system. Vitamin D3 deficiency is associated with cardiac autonomic imbalance. Administration of vitamin D3 in vitamin D deficient Parkinson's patient may may improve cardiac autonomic nerve function that can be interpreted by HRV.

ELIGIBILITY:
IInclusion criteria:

* Male patients with of Parkinson's disease diagnosed by neurologist with unilateral or bilateral involvement and mild to moderate disability according to Hoehn and Yahr (H-Y) scale (I-III)
* Age: 51-70 years
* BMI: 18.5-24.9 kg/m2
* Vitamin D3 deficient or insufficient
* On Levodopa medication

Exclusion criteria:

1. Patients with a history of drug abuse including alcoholism.
2. Patients on following drugs will be excluded-

   * Antioxidant vitamin supplements
   * Lipid lowering medications
   * Antihypertensive drug
   * Anti-arrhythmic drug
   * Sedatives
3. All patients with the history of or clinical manifestation of currently suffering from following diseases & condition will be excluded

   * Severe Cardiovascular disorders
   * Severe neurological disorders
   * Severe Respiratory disorders
   * Severe Renal insufficiency (S. Creatinine > 1.5 mg/dl, Acute or chronic kidney disease)
   * Severe Endocrine disease
   * Severe Arthritis
   * Severe Liver diseases
   * Severe Neoplastic disease
   * Severe Psychiatric disorder
   * Current use of iron, zinc, calcium, magnesium and multivitamin supplementation
   * Already performing yoga or breathing exercise
   * Hypercalcemia

Ages: 51 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Vitamin D3 supplementation has effect on cardiac autonomic nerve function in male Parkinson's disease patient | 8 weeks
  Altered cardiac autonomic nerve function

CONTACTS AND LOCATIONS:
Locations (1):
- Bangladesh Medical University, Dhaka, Shahbag, Bangladesh

IPD SHARING:
Plan to Share IPD: No